CLINICAL TRIAL: NCT06139861
Title: A Confirmatory Efficacy Trial of Engaging a Novel Sleep/Circadian Rhythm Target as Treatment for Depression in Adolescents
Brief Title: Better Sleep Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH129558-01A1 (NIH); R01MH129558-01A1 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Depression in Adolescence; Delayed Sleep Phase
Keywords: Depression; Adolescents; Sleep; Intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TranS-C (Experimental)
  Interventions: Behavioral: TranS-C
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: TranS-C — Transdiagnostic Sleep and Circadian Intervention (TranS-C) is an evidence based cognitive-behavioral sleep therapy.
  Arms: TranS-C
Behavioral: Psychoeducation — The overarching principle is to provide information about how sleep, stress, diet, health, exercise, accidents and mood are inter-related and have reciprocal effects.
  Arms: Psychoeducation

SUMMARY:
The overall aim of this proposal is a confirmatory efficacy trial sufficiently powered and designed to test the hypothesis that improving the relationship between biological circadian timing and waketime, a novel modifiable target, improves depression outcomes in a subgroup of adolescents with depression and a misaligned relationship between biological circadian timing and waketime utilizing a cognitive-behavioral sleep intervention.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* mental health/behavioral symptoms that would preclude productive engagement in study assessments or intervention (e.g., active psychosis; Bipolar Disorder; drug dependence
* severe or unstable medical or psychiatric condition such that treatment has changed within the last month or is expected to change during the course of the study or that would preclude ability to adhere to study procedures (e.g. terminal end-stage cancer)
* current use of medications or herbs with known effects on sleep
* plan to undergo or have had medication change in the last 8 weeks

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in phase angle difference (PAD) between DLMO and waketime (PADDLMO WAKETIME ) | baseline to end of treatment (0 and 2 months)
  Validated biological and behavioral assessment; range between 0 and 11 hours, with shorter numbers indicating worse alignment between circadian biology and behavior
Change in Children's Depression Rating Scale (CDRS-R) | baseline to end of treatment (anticipated average exposure 2 months), months 8 and 14
  Validated clinician administered depression symptom severity scale; range between 17 and 133, with higher numbers indicative of greater depression severity

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No